CLINICAL TRIAL: NCT06640465
Title: A Randomized, Placebo-Controlled Trial Comparing the Effects of Commercially Available Dietary Supplements on CoQ10 Concentrations
Brief Title: Comparing the Effects of Commercially Available Dietary Supplements on CoQ10 Concentrations
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: OvationLab (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: OvationLab
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Wellness; Health
Keywords: Coenzyme Q10; CoQ10; Geranylgeraniol; GG; Ubiquinol; Ubiquinone
MeSH Terms: interventions — ubiquinol; geranylgeraniol; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Ubiquinol + geranylgeraniol combination (Designs for Health - CoQnol™ 200) (Experimental)
  Interventions: Dietary Supplement: Ubiquinol + geranylgeraniol
- Geranylgeraniol (Annatto-GG™ 300) (Experimental)
  Interventions: Dietary Supplement: Geranylgeraniol
- Ubiquinol (Jarrow Formulas QH-absorb® 200 mg) (Experimental)
  Interventions: Dietary Supplement: Ubiquinol
- Ubiquinone (NOW CoQ10 200mg) (Experimental)
  Interventions: Dietary Supplement: Ubiquinone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ubiquinol + geranylgeraniol — Combination of ubiquinol and geranylgeraniol
  Arms: Ubiquinol + geranylgeraniol combination (Designs for Health - CoQnol™ 200)
Dietary Supplement: Geranylgeraniol — Geranylgeraniol alone
  Arms: Geranylgeraniol (Annatto-GG™ 300)
Dietary Supplement: Ubiquinol — Ubiquinol alone
  Arms: Ubiquinol (Jarrow Formulas QH-absorb® 200 mg)
Dietary Supplement: Ubiquinone — Ubiquinone alone
  Arms: Ubiquinone (NOW CoQ10 200mg)
Other: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to compare the safety and effectiveness of commercially available dietary supplements believed to increase coenzyme Q10 (CoQ10) concentrations.

An 8-week, randomized, placebo-controlled clinical trial will be conducted comparing the effectiveness of four commercially available dietary supplements on increasing CoQ10 concentrations and self-reported health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males or females age ≥ 40 years
2. Ability to read and speak English

Exclusion Criteria:

1. Daily use within the past 2 months of any dietary supplements containing CoQ10 or geranylgeraniol (GG)
2. Taking a statin medication within the past 6 months
3. Current daily usage of H2 blockers or PPI medications
4. Current daily use of bisphosphonates
5. Current daily tobacco smoker
6. Known allergies to any substance in the study products
7. Currently pregnant or lactating women or women planning to become pregnant in the next 12 weeks
8. Current diagnosis of a chronic health condition (e.g., cancer, Crohn's disease) deemed clinically contraindicated for the study protocol.
9. Participant in a clinical trial in the previous 30 days.
10. Participants unable to provide consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Plasma Coenzyme Q10 | Baseline and 8 weeks

SECONDARY OUTCOMES:
Comprehensive metabolic panel | Baseline and 8 weeks
  Alanine aminotransferase (ALT) in units per liter (U/L)
Lipid panel | Baseline and 8 weeks
  Low-density lipoprotein (LDL) in milligrams per deciliter (mg/dL)
Patient-Reported Outcomes Measurement Information System (PROMIS) - Global Health | Baseline and 8 weeks
  Raw scores range from 4 to 20, with higher scores indicating better global physical or mental health compared to the average
Profile of Mood States - Vigor Subscale | Baseline and 8 weeks
  Scores range from 0 to 32, with higher scores indicating better energy levels
Short Form 36 (SF-36) - Vitality Subscale | Baseline and 8 weeks
  Scores range from 0 to 100, with higher scores indicating greater vitality

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - True Health Center for Precision Medicine, El Dorado Hills, California
  - Cornerstone Health Community, Centennial, Colorado
  - CTMD Research, Palm Springs, Florida
  - Functional Medicine of Idaho, Eagle, Idaho
  - New Dawn Wellness and Medical Center, Houston, Texas
  - Vida Integrated Health, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and supporting information will be available within 6 months after the completion of the study.